CLINICAL TRIAL: NCT02780011
Title: A Phase I Study of the Combination of Alsertib (MLN8237) and Brentuximab Vedotin in Relapsed/Refractory CD30-Positive Lymphomas and Solid Malignancies
Brief Title: Alsertib (MLN8237) and Brentuximab Vedotin for Relapsed/Refractory CD30-Positive Lymphomas and Solid Malignancies
Acronym: AD3LE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Eric Bernicker, MD (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Eric Bernicker, MD, Study Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012815
Record Dates: First submitted 2016-02-24; First posted 2016-05-23 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: CD30-positive Lymphoma; CD30-positive Solid Tumor
Keywords: CD30+; Relapsed; Refractory; ALCL
MeSH Terms: conditions — Recurrence | interventions — Brentuximab Vedotin; MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alsertib and Brentuximab Vedotin (Experimental): Brentuximab vedotin at a fixed dose of 1.8 mg/kg will be administered by intravenous infusion on day 1 of every 21-day cycle. MLN8237 at a dose of 60 mg will be orally administered daily in 2 divided doses (30 mg qAM, 30 mg qPM) from days 1 to 7 of each 21-day cycle. MLN8237 dose will be escalated in 20-mg increments to the maximum dose of 100 mg (Level 2) or de-escalated in a 20-mg decrement to the minimum dose of 40 mg (Level -1).
  Interventions: Drug: Brentuximab Vedotin; Drug: Alsertib

INTERVENTIONS:
Drug: Brentuximab Vedotin — Antibody-drug conjugate composed of the anti-CD30 chimeric immunoglobulin G1 monoclonal antibody cAC10 and the antimicrotubule drug monomethyl auristatin E connected by a protease-cleavable linker.
  Other Names: Adcetris
Drug: Alsertib — Aurora A kinase inhibitor
  Other Names: MLN8237

SUMMARY:
This is an open label phase I trial designed to evaluate the maximum tolerated dose, dose-limiting toxicities, pharmacokinetics, and activity of the combination of alsertib (MLN8237) and brentuximab vedotin in patients with relapsed/refractory CD30-positive lymphomas and solid malignancies. Cohorts of 3-6 patients will receive escalating or de-escalating doses of MLN8237 based on a 3 + 3 design.

DETAILED DESCRIPTION:
This is an investigator-initiated, open label phase I trial designed to evaluate the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), pharmacokinetics, and activity of brentuximab vedotin in combination with MLN8237 in patients with relapsed/refractory CD30-positive lymphomas and solid malignancies.

Brentuximab vedotin at a fixed dose of 1.8 mg/kg will be administered on Day 1 every three weeks as a 30-minute outpatient intravenous infusion. MLN8237 will be orally administered in two divided doses from Days 1-7. The starting dose (level 0) of MLN8237 will be 60 mg daily given in two divided doses (30 mg qAM, 30 mg qPM).The dose of MLN8237 will be escalated in 20-mg increments up to 100 mg daily and de-escalated in 20-mg decrements to 40 mg daily. The fixed dose of brentuximab vedotin on Day 1 and daily dose of MLN8237 on Day 1-7 will constitute one treatment cycle. If no DLTs are observed in the last study cohort, the cohort will be expanded to include a total of 12 patients. If a de-escalation dose is required because 2 or more patients experience DLTs, the next lower cohort will be studied. If 2 or more patients do not experience DLTs, this dose will be declared the MTD. This cohort will be expanded to include 12 patients in order to study the biological endpoints and clinical benefit of the combination. If at any point during the expansion cohort phase of the trial 33% or more of the patients treated at the MTD/maximum administered dose experience a DLT, accrual of additional patients at this does level will cease and the next lowest dose may be explored.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care;
* Relapsed or refractory CD30-positive lymphoma such as Hodgkin's and anaplastic large cell lymphoma or CD30-positive cancer such as testicular embryonal carcinoma, cutaneous angiosarcoma, and nasopharyngeal non-keratinizing carcinoma or any CD30-positive solid tumor. CD30 positivity is defined as ≥ 25% CD30 expression by immunohistochemistry. (CD30 analysis will be performed by an in-house CLIA and CAP-accredited laboratory);
* Male or female patients aged ≥ 18 years;
* Adequate cardiac function (cardiac ejection fraction of ≥ 45%);
* Patients must have received at least two prior therapies for CD30-positive lymphoma or solid malignancy;
* Absolute neutrophil count > 1500/mm³, platelets > 100,000/mm³, and hemoglobin > 8 g/dL. Values must be obtained without the need for myeloid growth factor or platelet transfusion support within 14 days of the first dose of the study treatment; however, erythrocyte growth factor is allowed as per the American Society of Clinical Oncology guidelines;
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) and aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 x ULN. AST and/or ALT may be up to 5 x ULN if liver metastases are present;
* Adequate renal function as defined by a serum creatinine of < 2.0 mg/dL and calculated creatinine clearance of ≥ 30 mL/minute;
* Eastern Cooperative Oncology Group performance status of 0 to 2;
* Female patients must be either:

  * post-menopausal for at least one year before the screening visit, or
  * surgically sterilized, or
  * willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study;
* Male patients, even if surgically sterilized (i.e., post-vasectomy status), must agree to use an acceptable contraceptive method during the course of the study and for 4 months after the last dose of alisertib.

Exclusion Criteria:

* Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%;
* Prior allogeneic bone marrow or organ transplantation;
* Expected survival of less than 4 weeks;
* Known gastrointestinal (GI) disease or GI procedures that could interfere with the oral absorption of or tolerance to alisertib. Examples include but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease;
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease;
* Known cerebral or meningeal disease (Hodgkin's lymphoma or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy;
* Symptomatic neurologic disease that compromises normal activities of daily living or requires medication;
* Requirement for constant or intermittent administration of a proton pump inhibitor, a H2 antagonist, or pancreatic enzymes. Intermittent use of antacids or H2 antagonists is allowed;
* Systemic infection requiring intravenous antibiotic therapy within 14 days preceding the first dose of the study treatment or other severe viral or bacterial infection;
* Absolute QT interval of > 460 msec in the presence of > 4.0 mEq/L potassium and > 1.8 mg/dL magnesium;
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiogram abnormality at screening has to be documented by the investigator as not medically relevant;
* Female patient who is pregnant or breastfeeding. Confirmation that the subject is not pregnant must be established by a negative serum beta human chorionic gonadotropin pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women;
* Patient has received other investigational drugs within 14 days of enrollment;
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study;
* Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study;
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy;
* Treatment with clinically significant enzyme inducers, such as phenytoin, carbamazepine, phenobarbital, rifampin, rifabutin, rifapentine, and St. John's wort, within 14 days prior to the first dose of alisertib;
* Known history of human immunodeficiency virus, hepatitis B, or hepatitis C infection. Testing is not required in the absence of clinical findings or suspicion;
* Prior administration of an Aurora A kinase-targeted agent, including alisertib;
* Prior administration of brentuximab vedotin is allowed only if the patient did not experience disease progression while on treatment;
* Known hypersensitivity to recombinant proteins, murine proteins, or any excipient contained in the drug formulation of brentuximab vedotin;
* Concurrent or recent (within 2 weeks) use of strong cytochrome P450 (CYP) 3A4 inhibitors such as ketoconazole, itraconazole, clarithromycin, atanazir, inddinavir, nefazodone, neflinavir, ritonavir, saquinavir, telithromycin, and voriconazole;
* Concurrent or recent (within 2 weeks) use of potent CYP3A4 inducers such as dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's wort;
* Concurrent or recent (within 2 weeks) use of a P-glycoprotein inhibitor such as cyclosporine, ketoconazole, ritonavir, saquinavir, tacrolimus, or verapamil;
* Receipt of corticosteroids within 7 days prior to the first dose of the study treatment, unless the patient has been taking a continuous dose of no more than 15 mg/day of prednisone for at least 1 month prior to the first dose of the study treatment. Low-dose steroid use for the control of nausea and vomiting will be allowed. Topical steroid use is permitted. Inhaled steroids are permitted;
* Inability to swallow oral medication or inability or unwillingness to comply with the administration requirements related to alisertib;
* Administration of myeloid growth factors or platelet transfusion within 14 days prior to the first dose of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Approximately 12 weeks
  Determine the MTD of the alsertib (MLN8237) and brentuximab vedotin combination in patients with relapsed/refractory CD30-positive lymphomas and solid malignancies.

SECONDARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Approximately 12 weeks
  Describe the DLTs and other toxicities associated with the alsertib (MLN8237) and brentuximab vedotin combination as assessed by CTCAE v4.0.
Recommended phase 2 dose (RP2D) | Approximately 12 weeks
  Determine the RP2D of the alsertib (MLN8237) and brentuximab vedotin combination.
Antitumor activity | Approximately 12 weeks
  Document the antitumor activity of the alsertib (MLN8237) and brentuximab vedotin combination as assessed by modified IWG criteria and RECIST 1.1.
Area under the plasma concentration versus time curve | Cycle 1, Day 1 at pre-infusion and 10 min, 24 h, and 48 h post-infusion; trough sample on Cycle 1, Day 8; and Cycle 2, Day 1 at pre-infusion and 12 h and 24 h post-infusion.
  Determine the area under the plasma concentration versus time curve of alsertib (MLN8237) and brentuximab vedotin.

OTHER OUTCOMES:
H3K activity | Approximately 12 weeks
  Measure H3K activity in peripheral blood mononuclear cells and tumor tissue following treatment with the combination of alsertib (MLN8237) and brentuximab vedotin.
Correlation between CD30 detection method and clinical response | Approximately 12 weeks
  Explore the correlation between CD30 detection method (aptamer-mediated flow cytometric detection vs. immunohistochemical detection) and clinical response to the combination of alsertib (MLN8237) and brentuximab vedotin.

CONTACTS AND LOCATIONS:
Overall Officials: Swami Padmanabhan Iyer, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and materials on human subjects will be shared with other eligible investigators through appropriate means in accordance with the NIH policy on Sharing Research Data (NIH Guide, February 26, 2003). Data will be also shared with the funding agency and regulatory agencies as required. Data will be shared with other investigators within the limits of HIPAA and other patient confidentiality requirements. This will generally require removal of all patient identifiers for all source documents and the use of arbitrarily assigned one-way identifiers. In some cases, requestors will be asked to sign a formal data sharing agreement that will provide for a commitment to use data only for research purposes and not to identify individuals, keep the data secure, and destroy or return data after analyses are complete. Prior approval will be obtained from collaborating investigators, research sponsors, and/or other stake-holders before sharing if proprietary information or products are involved.